CLINICAL TRIAL: NCT00636285
Title: Phase 1, Open-Label, Dose-Ranging, Safety and Pharmacokinetics Study in Adults of BSYX-A110, a Human Chimeric Anti-Staphylococcal Monoclonal Antibody for the Prevention of S. Epidermidis Infection in Low Birth Weight Infants
Brief Title: Safety and Pharmacokinetics Study in Adults for the Prevention of S. Epidermidis Infection in Low Birth Weight Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosynexus Incorporated (Industry)
Responsible Party: Gerald Fischer, MD, President and CEO, Biosynexus Incorporated
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MAB-A001
Record Dates: First submitted 2008-02-27; First posted 2008-03-14 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-10

CONDITIONS: Staphylococcal Sepsis
Keywords: A110; Safety
MeSH Terms: interventions — pagibaximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 2 (Experimental): BSYX-A110, Dosed intravenously, 3mg/kg
  Interventions: Drug: BSYX-A110
- 3 (Experimental): BSYX-A110, Dosed intravenously, 10mg/kg
  Interventions: Drug: BSYX-A110

INTERVENTIONS:
Drug: Placebo — Placebo
  Other Names: Pagibaximab; BSYX-A110
  Arms: 1
Drug: BSYX-A110 — BSYX-A110, Dosed intravenously, 3 mg/kg
  Other Names: Pagibaximab
  Arms: 2
Drug: BSYX-A110 — BSYX-A110, Dosed intravenously, 10 mg/kg
  Other Names: Pagibaximab
  Arms: 3

SUMMARY:
The purpose of this Phase 1 study is to evaluate the safety and pharmacokinetics of BSYX-A110 in a small number of healthy adult volunteers. Following the demonstration of safety in adults, this anti-Staphylococcal monoclonal antibody will then be evaluated in the target population of hospitalized low birth weight neonates.

DETAILED DESCRIPTION:
This study will evaluate the safety of three doses of BSYX-A110 in adults before initiating studies in the target population of low birth weight infants. This will be an open label, dose-ranging study of BSYX-A110 in 12 adults. The dose levels to be evaluated are 3, 10 and 20 mg/kg. Each dose level will enroll 4 adult volunteers who will receive one dose of BSYX-A110 intravenously. The primary endpoint of this study is safety and tolerability. The secondary endpoints include the pharmacokinetics of the rise in anti-LTA antibody and opsonic activity against S. epidermidis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 18 years of age or older.
2. Subjects must in good general health, without significant medical history, physical examination findings or clinical laboratory abnormalities.
3. Negative screening pre-treatment pregnancy test for female subjects.
4. Subjects of childbearing potential must agree to use an acceptable method of contraception throughout the course of the study.
5. All aspects of the protocol explained and written informed consent obtained.

Exclusion Criteria:

1. Known or suspected immunodeficiency (e.g. HIV infection, significant risk factors for HIV, primary immunosuppressive disorder), use of immunosuppressive or antineoplastic drugs except corticosteroids used for indications other than immunosuppression.
2. Clinically significant laboratory abnormality (greater than 1.5 upper limit of normal.).
3. Serology positive for HIV, hepatitis B surface antigen or hepatitis C antibody.
4. History of leukemia, lymphoma or other malignancy.
5. Clinically significant cardiac, respiratory, renal, hepatic, neurological disorder
6. Pregnant or lactating females (women of childbearing potential will undergo a pregnancy test).
7. Receipt of any vaccine within 30 days.
8. History of drug or alcohol dependence, or significant acute or chronic medical or psychiatric illness which would limit the subject's ability to complete the study and/or compromise the objectives of the study.
9. Fever or acute illness within 3 days prior to treatment. (These subjects can be rescheduled for treatment at a later date).
10. Participation in another investigational drug or vaccine trial within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2001-04; Primary Completion 2001-09 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability. | 28 days

SECONDARY OUTCOMES:
To evaluate the serum levels (pharmacokinetics) of anti-LTA antibodies (ELISA; the functional opsonic activity against S. epidermidis; and correlate the levels of anti-LTA antibodies achieved with opsonic activity against S. epidermidis | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Weisman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- See also: Biosynexus Incorporated — http://www.biosynexus.com